CLINICAL TRIAL: NCT05114109
Title: Isatuximab in Type I Cryoglobulinemia: A Prospective Pilot Study
Brief Title: Isatuximab in Type I Cryoglobulinemia
Acronym: ICE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-001992-17
Record Dates: First submitted 2021-09-27; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-09

CONDITIONS: Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Cryoglobulinemic Vasculitis
MeSH Terms: conditions — Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Cryoglobulinemia, Familial Mixed | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isatuximab (Experimental): Isatuximab will be given intravenously.
  Interventions: Drug: Isatuximab Injection

INTERVENTIONS:
Drug: Isatuximab Injection — Isatuximab will be given intravenously at 10mg/kg at day 0, week (W)1, W2, W3, and W4 then every 2 weeks for a total of 12 infusions.

SUMMARY:
Cryoglobulinaemia is defined as the presence of immunoglobulins in the serum, which reversibly precipitate and form a gel when the temperature drops below 37°C and redissolve upon re-warming. Classification includes three subgroups based on Immunoglobulin (Ig) composition. Type I cryoglobulinaemia consists of only one isotype or subclass of immunoglobulin. Types II and III are classified as mixed cryoglobulinaemia (MC) because they include both IgG and IgM components. Overall, cryoglobulinaemia is considered a rare disease (<5/10,000 in the general European and North American population), although prevalence is likely to be higher in some areas such as the Mediterranean Basin. MC vasculitis is a multi-organic disease involving kidneys, joints, skin, and peripheral nerves. In type I cryoglobulinaemic vasculitis, searching for an underlying plasma-cell neoplasms is mandatory. Cryoglobulinaemia composed of IgG is more often found in multiple myeloma or monoclonal gammapathy of unknown significance. The course of MC vasculitis varies widely, and the prognosis is influenced by both MC-induced damage to vital organs and co-morbidities associated with underlying diseases. Type I cryoglobulinaemic vasculitis is a plasma cell associated disorder at the crossroad between autoimmunity and plasma-cell neoplasm. Treatment should be modulated according to the underlying associated disease and the severity of internal organ involvement. The overall 10-year survival after a diagnosis of cryoglobulinaemic syndrome ranges from 50% to 90% in case of renal involvement. The main therapeutic goal must be the cure of the underlying haematological disease (overwhelmingly plasma-cell neoplasms). The most common neoplasias are multiple myeloma (predominantly associated with type I cryoglobulinaemia and hyper-viscosity) in more than 50% of cases. Treating the underlying monoclonal disorder has been associated with improvement/stabilization of cryoglobulinaemic symptoms in most patients with type I cryoglobulinemia, although negativation of serum cryoglobulins was achieved in only half the patients. Alkylating agents and bortezomib are the main therapeutic options, but are associated with side effects including neuropathy. Patients presenting with symptomatic hyperviscosity require urgent therapeutic intervention using plasma exchange or plasmapheresis to remove cryoglobulins from the circulation. There is no standard of care or international guidelines for treatment of type 1 cryoglobulinemia. Isatuximab is an anti-CD38 monoclonal antibody that has been effective to treat relapsed or refractory multiple myeloma. Autoreactive plasma cells represent a key player in autoimmune disorders and particularly in type I cryoglobulinemia. Type I cryoglobulinemia is a model of plasma cell associated disorder at the crossroad between autoimmunity and plasma-cell neoplasm. However, rituximab fails to target this population and is poorly effective in this condition. Thus, there is an unmeet need for plasma cell targeted therapy in type I cryoglobulinemia. Clonal plasma cells in type I cryoglobulinemia do express surface CD38, providing a rationale for the use of isatuximab in cryoglobulinemia. Although the biology of the clonal plasma cell in type I cryoglobulinemia is distinct from that of Amyloid light-chain (AL) amyloidosis, they are models of hematological diseases associated with monoclonal Ig and whose tumor mass is low. In AL amyloidosis anti-CD38 targeted therapy was highly efficient as monotherapy in treatment naïve patients and relapsers. Thus, Isatuximab represents a highly promising therapy in type I cryoglobulinemia that could be use as monotherapy.

This study is a Phase 2 pilot prospective study of 21 patients with type I cryoglobulinemia treated by Isatuximab. Isatuximab will be given intravenously at 10 mg/kg at day 0, week (W)1, W2, W3, and W4 then every 2 weeks for a total of 12 infusions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Written informed consent
* Indolent Multiple myeloma or monoclonal gammopathy of unknown significance (MGUS) with monoclonal IgG component
* Active cryoglobulinemia vasculitis defined by positive type I IgG cryoglobulinemia and a clinically active cryoglobulinemia with skin, joint, renal, and/or peripheral involvement,
* Treated naïve or relapsers type I cryoglobulinemia patients
* Affiliated to National French social security system
* Contraception :

  1. Male participants : A male participant must agree to use a highly effective method of contraception during the participation period and for at least 5 months after the last dose of study treatment and refrain from donating sperm during this period.
  2. Female participants : A female participant is eligible to participate if she is not pregnant, not breastfeeding, and with at least one of the following conditions:
* Not a female of childbearing potential (FCBP), OR
* A FCBP who must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 24 hours of starting study medication and must apply a highly effective method of contraception during the participation period and for at least 5 months after the last dose of study treatment and refrain from donating oocyte during this period
* HIV negative serology; negative HBs Ag test; HCV negative serology and/or negative HCV RNA if positive HCV serology

Exclusion Criteria:

* Patient with a vasculitis unrelated to cryoglobulinemia
* Patient with non-active cryoglobulinemia vasculitis,
* Patient with diagnosis of multiple myeloma
* Patient treated with immunosuppressant (e.g alkylating agent, Rituximab, chemotherapy for plasma-cell neoplasms) introduced or increased in the month prior to the inclusion,
* Live vaccines within 30 days prior to baseline or concurrently with Isatuximab
* Infection requiring hospitalization and/or use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within 60 days of Day 0.
* Active tuberculosis
* HIV positive, positive Ag HbS, positive HCV RNA
* Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose excessive risk to the patient or may interfere with compliance or interpretation of the study results.
* Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study therapy that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
* Hypersensitivity to the active substances (isatuximab and premedication) or to any of their excipients
* Received any investigational drug within 14 days prior to inclusion or within 5 half-lives of the investigational drug, whichever is longer.
* Participation in another interventional study or being in the exclusion period at the end of a previous study.
* Vulnerable populations

  * pregnant or breastfeeding women
  * Persons deprived of liberty by judicial or administrative decision
  * Persons under psychiatric care without their consent
  * Adults subject to a legal protection measure
  * Persons unable to express their consent
* Neutrophils < 1000/mm3
* Platelets < 75000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response W20 | 20 Weeks
  Complete clinical response rate of cryoglobulinemia vasculitis symptoms. The complete clinical response is defined by the remission of all affected organs involved at baseline and the absence of clinical relapse according to the international guidelines.
  * The skin and articular remissions are evaluated clinically (disappearance of purpura and/or ulcers, disappearance of arthritis).
  * Renal remission is evaluated biologically (proteinuria <0.5g/24h or proteinuria/creatinuria <50 mg/mmol).
  * Neurological remission is evaluated clinically (any improvement of pains and paresthesia by visual analogue scales, any improvement of muscular testing in case of motor impairment at baseline) and electrophysiologically (improvement of electromyogram abnormalities compared to baseline).

SECONDARY OUTCOMES:
Adverse event | 20 Weeks
  Frequency and severity of adverse clinical events
Response | 12 and 20 weeks
  Complete, partial and non-clinical response rates
Remission BVAS | 12 and 20 weeks
  Rate of patients remaining in remission with a Birmingham Vasculitis Activity Score (BVAS), BVAS=0
Early failures | 4 weeks
  Rate of early failures (non-clinical response)
Cryoglobulinemia | 12 and 20 weeks
  Rate of cryoglobulinemia clearance
Rheumatoid factor | 12 and 20 weeks
  Rate of negativation of rheumatoid factor activity
C4 complement | 12 and 20 weeks
  Rate of normalization of C4 complement level
Renal complete remission | 12 and 20 weeks
  Rate of renal complete remission defined as proteinuria <0.5g/24h or proteinuria/creatinuria <50 mg/mmol, disappearance of hematuria, and glomerular filtration rate ≥60ml/min/1.73m²
Clinical relapse | 20 weeks
  Clinical relapse rate defined by de novo appearance or reappearance of a manifestation attributable to cryoglobulinemia vasculitis
Relapse | 48 weeks
  Incidence of relapse
Gammaglobulin | 20 weeks
  Mean change of gammaglobulin level from baseline to Week 20
CD19+ B cells | 20 weeks
  Mean change of CD19+ B cells level from baseline to Week 20
Quality of life SF36 | 20 weeks
  Quality of life assessed by the mean variation of the Short Form 36 Health Survey Questionnaire (SF-36) from baseline to Week 20 The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Infections | 48 weeks
  Rate of infections

IPD SHARING:
Plan to Share IPD: Undecided